CLINICAL TRIAL: NCT00799994
Title: Effect of Acutely Lowering Intraocular Pressure on Multifocal Visual Evoked Potential Testing
Brief Title: Does Lowering Eye Pressure Affect the Results Obtained From Objective Visual Field Testing?
Status: Completed | Type: Observational
Sponsor: Wills Eye (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, L. Jay Katz MD, Glaucoma Service Chief, Wills Eye
Other Study IDs: 04-653
Record Dates: First submitted 2008-11-28; First posted 2008-12-01 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-11

CONDITIONS: Glaucoma
Keywords: glaucoma; intraocular pressure; multifocal visually evoked potentials
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Patients that have medical intervention in an attempt to lower intraocular pressure (oral or topical)
- 2: Patients who have received no intervention

SUMMARY:
A study to determine whether a patient's range of vision test results improve after their eye pressure is lowered by 30% or more by testing on a new machine called the Accumap and how to learn how much the Accumap's results change from one test to another within the same person.

The investigators believe that Multifocal VEP readings (Accumap)(and therefore visual function and ganglion cell function) improve after acutely lowering intraocular pressure.

DETAILED DESCRIPTION:
Accumap testing will be performed before and two to three hours after treatment is initiated to lower IOP. In eye that have bilateral treatment, one eye will be assigned randomly to the study. The mean multifocal objective perimetry amplitude will be compared before and after IOP reduction. Also, the mean amplitudes of five circumferential zones will be compared before and after IOP lowering. Visual field testing and HRT testing will be performed before and after treatment as well if possible. Paired t-tests will be performed no pre-and post-treatment mean MOP amplitude values and circumferential zones to determine statistical significance. A second group of patients whose pressures will not be lowered will also be tested with Accumap at baseline and two hours afterwards, in order to examine reproducibility of mean MOP amplitude and mean circumferential amplitude. HVF and HRT testing will also be obtained on thes patients when possible.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients seen that have their intraocular pressures lowered by at least 30% over the course of two hours.

Exclusion Criteria:

* Recent (within 6 weeks) intraocular surgery
* Visual acuity worse than 20/40
* Pathology unrelated to glaucoma (retinal disease, stroke, brain tumor, etc) associated with visual field defect
* Prior corneal transplant, corneal edema, or corneal diseases such as keratoconus or dense scarring

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: glaucoma service
Sampling Method: Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2004-10; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
lowering of intraocular pressure will cause an acute improvement in MfVEP (multifocal visually evoked potential) amplitude readings | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: L. Jay Katz, MD, Principal Investigator — Wills Eye Institute
Locations (1):
- Wills Eye, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No